CLINICAL TRIAL: NCT00332995
Title: Double-blind, Randomized, Placebo Controlled Trial to Study Safety, Local and Systemic Availability of TMC120 From a Vaginal Ring.
Brief Title: Safety and Feasibility Study of Dapivirine (TMC120) Vaginal Ring in Belgium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Zeda Rosenberg ScD, International Partnership for Microbicides
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM008, TMC120-C131
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Contraceptive Devices, Female

INTERVENTIONS:
Drug: dapivirine (TMC120) vaginal ring

SUMMARY:
This Phase I trial will assess the feasibility of using a vaginal ring to deliver the candidate microbicide dapivirine (TMC120) for 7 days. The study population will consist of 13 healthy, sexually abstinent women. Safety and tolerability will be assessed through clinical and laboratory assessments. Feasibility of drug delivery will be assessed by measuring dapivirine (TMC120) concentrations in vaginal fluids, vaginal and cervical epithelial tissue, and plasma.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-50 years
* Willing and able to provide written informed consent
* HIV-uninfected and otherwise healthy
* Willing to abstain from sexual activity and from use of vaginal products while participating in the study
* Currently using oral contraceptives for pregnancy prevention
* Willing to use oral contraceptives as needed to avoid menstruation while taking part in this study

Exclusion Criteria:

* History of allergy to TMC120 or to the constituents of the vaginal ring
* History of diagnosis of and/or treatment for a sexually transmitted disease within the last three months
* History of genital tract surgery within the last month
* Currently pregnant or breastfeeding, or within two months of last pregnancy outcome
* Currently or within one month of participating in any other clinical research study
* Current vulvar or vaginal symptoms / abnormalities that could influence the study results
* Current non-iatrogenic pelvic/colposcopic exam findings involving deep epithelial disruption
* Current diagnosis of any genital infection
* Smoking more than 10 cigarettes / day

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13
Dates: Start 2005-07; Study Completion 2005-08

PRIMARY OUTCOMES:
Safety and tolerability of seven-day use of a vaginal ring containing dapivirine (TMC120).
Assess dapivirine (TMC120) concentrations in vaginal fluids, vaginal and cervical epithelial tissue, and plasma during and after seven-day use of a vaginal ring containing dapivirine (TMC120).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Luc Van Bortel, Principal Investigator — University Ghent
Locations (1):
- Drug Research Unit Gent, Ghent, Belgium